CLINICAL TRIAL: NCT06393712
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacodynamics of Intrathecally Administered ALN-APP in Patients With Cerebral Amyloid Angiopathy (CAA)
Brief Title: A Phase 2 Trial of ALN-APP in Patients With Cerebral Amyloid Angiopathy
Acronym: cAPPricorn-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-APP-002; 2023-510137-29-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-19; First posted 2024-05-01 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Amyloid Angiopathy
Keywords: CAA
MeSH Terms: conditions — Cerebral Amyloid Angiopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALN-APP (Experimental): Participants will be administered multiple doses of ALN-APP during the double-blind treatment period and optional open-label extension period.
  Interventions: Drug: ALN-APP
- Placebo/ALN-APP (Placebo Comparator): Participants will be administered multiple doses of placebo during the double-blind treatment period. Participants who continue into the optional open-label extension period will be administered multiple doses of ALN-APP.
  Interventions: Drug: Placebo; Drug: ALN-APP

INTERVENTIONS:
Drug: Placebo — Placebo will be administered intrathecally
  Arms: Placebo/ALN-APP
Drug: ALN-APP — ALN-APP will be administered intrathecally
  Other Names: mivelsiran

SUMMARY:
The purpose of the study is to evaluate the effect of ALN-APP on measures of CAA disease progression and to characterize the safety, tolerability, and pharmacodynamics (PD) of ALN-APP in adult patients with sporadic CAA (sCAA) and Dutch-type CAA (D-CAA). The study will be conducted over 2 periods: a 24-month double-blind treatment period and an optional 18-month open-label extension (OLE) period. The estimated duration of study participation, inclusive of screening, treatment, and additional safety follow-up, is up to 50 months.

ELIGIBILITY:
Inclusion Criteria (sporadic CAA patients):

* Is 50 years or older
* Has probable CAA per the Boston Criteria Version 2.0

Inclusion Criteria (Dutch-type CAA patients):

* Is 30 years or older
* Has known E693Q amyloid precursor protein (APP) gene mutation for Dutch-type CAA

Exclusion Criteria:

* Moderate or severe stage Alzheimer's disease (AD) or significant cognitive impairment (CI)
* Has a history of previous clinical intracerebral hemorrhage (ICH) with onset less than 90 days prior to anticipated randomization in the study
* Has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3×upper limit of normal (ULN) at Screening
* Has estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m^2 at Screening
* Has recently received an investigational agent
* Has had treatment with amyloid-targeting antibody

Note: other protocol defined inclusion / exclusion criteria apply

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Double-blind Treatment Period: Annualized Rate of New Lobar Cerebral Microbleeds (CMBs) Assessed on Magnetic Resonance Imaging (MRI) of Brain in Patients with Sporadic Cerebral Amyloid Angiopathy (sCAA) | Up to 24 months

SECONDARY OUTCOMES:
Double-blind Treatment Period: Global Rank Based on Severity, Count, Symptom Burden, and Timing of New Clinical Hemorrhagic Events and Hemorrhagic Lesions Assessed on MRI of Brain | Up to 24 months
Double-blind Treatment Period: Change from Baseline Over Time in Cerebrovascular Vasoreactivity Measured by Blood Oxygenation Level Dependent (BOLD) Parameters with Visual-evoked Functional MRI | Up to 24 months
Double-blind Treatment Period: Incidence of New Cerebral Hemorrhagic Lesions and White Matter Hyperintensities Assessed on MRI of Brain | Up to 24 months
Double-blind Treatment Period: Change from Baseline Over Time in the Total Cerebral Amyloid Angiopathy (CAA) Small Vessel Disease Score Assessed on MRI of Brain | Up to 24 months
Double-blind Treatment Period: Change from Baseline in Soluble Amyloid Precursor Protein Alpha (sAPPα) Concentration in Cerebrospinal Fluid (CSF) | Up to 24 months
Double-blind Treatment Period: Change from Baseline in Soluble Amyloid Precursor Protein Beta (sAPPβ) Concentration in CSF | Up to 24 months
Double-blind Treatment Period and Open-label Extension (OLE) Period: Frequency of Adverse Events | Up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (38):
- United States (21):
  - Clinical Trial Site, Palo Alto, California
  - Clinical Trial Site, Sacramento, California
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, Gainesville, Florida
  - Clinical Trial Site, Jacksonville, Florida
  - Clinical Trial Site, Naples, Florida
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Lexington, Kentucky
  - Clinical Trial Site, New Orleans, Louisiana
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Plymouth, Massachusetts
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Canton, Ohio
  - Clinical Trial Site, Cleveland, Ohio
  - Clinical Trial Site, Abington, Pennsylvania
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, Seattle, Washington
- Australia (5):
  - Clinical Trial Site, Brisbane, Queensland
  - Clinical Trial Site, Adelaide, South Australia
  - Clinical Trial Site, Heidelberg, Victoria
  - Clinical Trial Site, Parkville, Victoria
  - Clinical Trial Site, Nedlands, Western Australia
- Canada (6):
  - Clinical Trial Site, Calgary, Alberta
  - Clinical Trial Site, Kelowna, British Columbia
  - Clinical Trial Site, Moncton, New Brunswick
  - Clinical Trial Site, Hamilton, Ontario
  - Clinical Trial Site, Ottawa, Ontario
  - Clinical Trial Site, Toronto, Ontario
- Netherlands (3):
  - Clinical Trial Site, Amsterdam
  - Clinical Trial Site, Leiden
  - Clinical Trial Site, Nijmegen
- Switzerland (2):
  - Clinical Trial Site, Bern
  - Clinical Trial Site, Geneva
- Clinical Trial Site, London, LND, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Access to data may be declined where there is likelihood a patient could be identified or other feasibility issue, where there is a potential conflict of interest, a planned business activities or an actual or potential competitive risk. Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Timeframes for data access may vary and can take up to 6 months or more.
  Requests for access to data can be submitted via the website www.vivli.org. Questions can also be directed to datasharing@alnylam.com.